CLINICAL TRIAL: NCT03033511
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of Rovalpituzumab Tesirine as Maintenance Therapy Following First-Line Platinum-Based Chemotherapy in Subjects With Extensive Stage Small Cell Lung Cancer (MERU)
Brief Title: A Study of Rovalpituzumab Tesirine as Maintenance Therapy Following First- Line Platinum-Based Chemotherapy in Participants With Extensive Stage Small Cell Lung Cancer (MERU)
Acronym: MERU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Independent Data Monitoring Committee recommendation
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-298; 2016-003503-64 (EudraCT Number)
Expanded Access: NCT03503890 (No longer available)
Record Dates: First submitted 2017-01-25; First posted 2017-01-26 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Small Cell Lung Cancer
Keywords: Extensive-Stage Small Cell Lung Cancer (ED SCLC); Cancer; Platinum-Based Chemotherapy; Rovalpituzumab tesirine; first-line chemotherapy; Small Cell Lung Cancer (SCLC); Delta-like protein 3 (DLL3)
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — Dexamethasone; rovalpituzumab tesirine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rovalpituzumab tesirine/dexamethasone (Experimental): Rovalpituzumab tesirine/dexamethasone every 6 weeks (q6 wk); omitting every third cycle
  Interventions: Drug: Rovalpituzumab tesirine; Drug: Dexamethasone
- Placebo (Experimental): Placebo q6 wk; omitting every third cycle
  Interventions: Drug: Placebo for dexamethasone; Drug: Placebo for rovalpituzumab tesirine

INTERVENTIONS:
Drug: Placebo for dexamethasone — Placebo for dexamethasone PO twice daily on Day -1, Day 1 (the day of dosing), and Day 2 of each 6 week cycle, omitting every third cycle.
  Arms: Placebo
Drug: Placebo for rovalpituzumab tesirine — Placebo for rovalpituzumab tesirine administered intravenously Day 1 of each 6-week cycle, omitting every third cycle
  Arms: Placebo
Drug: Rovalpituzumab tesirine — Rovalpituzumab tesirine 0.3 mg/kg administered intravenously Day 1 of each 6-week cycle, omitting every third cycle
  Arms: Rovalpituzumab tesirine/dexamethasone
Drug: Dexamethasone — Dexamethasone 8 mg administered orally (PO) twice daily on Day -1, Day 1 (the day of dosing), and Day 2 of each 6 week cycle, omitting every third cycle.
  Arms: Rovalpituzumab tesirine/dexamethasone

SUMMARY:
This is a Phase 3, randomized, double-blind, placebo-controlled, multinational, and multicenter study to evaluate the efficacy of rovalpituzumab tesirine as maintenance therapy following first-line platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive-stage disease small cell lung cancer (ED SCLC) at initial diagnosis with ongoing clinical benefit (stable disease [SD], partial response [PR], or complete response [CR]) following completion of 4 cycles of first-line platinum-based therapy
* Participant is eligible to be randomized at least 3 but no more than 9 weeks from Day 1 of the fourth cycle of first-line platinum-based chemotherapy.
* Participants with a history of central nervous system (CNS) metastases prior to the initiation of first-line platinum-based chemotherapy must have received definitive local treatment and have documentation of stable or improved CNS disease status
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
* Participants must have adequate bone marrow, renal and hepatic function
* Availability of archived or representative tumor material for assessment of DLL3 expression

Exclusion Criteria:

* Any prior systemic chemotherapy, small molecule inhibitors, immune checkpoint inhibitors, other monoclonal antibodies, antibody-drug conjugates, radioimmunoconjugates, T-cell or other cell-based or biologic therapies, or any other anti-cancer therapy than that described in inclusion criteria for SCLC.
* Any disease-directed radiotherapy (except prophylactic cranial irradiation, palliative radiotherapy to a radiographically documented non-progressing lesion for symptom control, or pre-planned radiotherapy for CNS metastases present prior to start of first-line therapy and non-progressing) after last dose of first-line chemotherapy.
* Prior exposure to a pyrrolobenzodiazepine (PBD-based) or indolinobenzodiazepine-based drug, prior participation in a rovalpituzumab tesirine clinical trial, or known hypersensitivity or other contraindications to rovalpituzumab tesirine or excipient contained in the drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (308):
- United States (54):
  - Clearview Cancer Institute /ID# 156699, Huntsville, Alabama
  - University of South Alabama /ID# 160975, Mobile, Alabama
  - Highlands Oncology Group /ID# 156722, Fayetteville, Arkansas
  - Marin Cancer Care /ID# 159207, Greenbrae, California
  - Ucsd /Id# 157764, La Jolla, California
  - LA Hem-Oncology Med Group /ID# 156717, Los Angeles, California
  - Palo Alto Veterans Institute for Research /ID# 203695, Palo Alto, California
  - St Jude Hospital dba St Joseph /ID# 156526, Santa Rosa, California
  - Icri /Id# 157765, Whittier, California
  - Kaiser Permanente Lone Tree /ID# 159331, Lone Tree, Colorado
  - Christiana Care Health Service /ID# 159212, Newark, Delaware
  - Holy Cross Hospital /ID# 156716, Fort Lauderdale, Florida
  - University of Florida - Archer /ID# 155799, Gainesville, Florida
  - Memorial Cancer Institute /ID# 156673, Hollywood, Florida
  - Memorial Cancer Institute /ID# 164052, Hollywood, Florida
  - Cancer Specialists of North Florida - Southpoint /ID# 156595, Jacksonville, Florida
  - Georgia Cancer Center /ID# 201894, Atlanta, Georgia
  - Southeastern Regional Medical /ID# 163064, Newnan, Georgia
  - St. Luke's Mountain States Tumor Institute - Boise /ID# 156691, Boise, Idaho
  - NorthShore University HealthSystem - Evanston Hospital /ID# 156664, Evanston, Illinois
  - Ingalls Memorial Hosp /ID# 156685, Harvey, Illinois
  - Goshen Center for Cancer Care /ID# 156682, Goshen, Indiana
  - Ashland-Bellefonte Cancer Ctr /ID# 202901, Ashland, Kentucky
  - University of Louisville /ID# 156683, Louisville, Kentucky
  - Ochsner Clinic Foundation /ID# 159136, Baton Rouge, Louisiana
  - Henry Ford Health System /ID# 156712, Detroit, Michigan
  - Sparrow Regional Cancer Center, Sparrow Health System /ID# 156590, Lansing, Michigan
  - Mayo Clinic - Rochester /ID# 160181, Rochester, Minnesota
  - MidAmerica Division, Inc. /ID# 163530, Kansas City, Missouri
  - Billings Clinic /ID# 201788, Billings, Montana
  - Nebraska Hematology Oncology /ID# 156534, Lincoln, Nebraska
  - MD Anderson Cancer Center at Cooper - Camden /ID# 156681, Camden, New Jersey
  - Northwell Health - Monter Cancer Center /ID# 159252, Lake Success, New York
  - Icahn School of Med Mt. Sinai /ID# 159210, New York, New York
  - Stony Brook University Hospital /ID# 159272, Stony Brook, New York
  - Montefiore Medical Center /ID# 201845, The Bronx, New York
  - Duke University Medical Center /ID# 156706, Durham, North Carolina
  - Cone Health /ID# 156689, Greensboro, North Carolina
  - Cone Health /ID# 163612, Greensboro, North Carolina
  - Eastern Carolina University /ID# 159264, Greenville, North Carolina
  - Gabrail Cancer Center Research /ID# 156667, Canton, Ohio
  - Kaiser Permanente, NW /ID# 201793, Portland, Oregon
  - Thomas Jefferson University /ID# 156719, Philadelphia, Pennsylvania
  - VA Pittsburgh HealthcareSystem /ID# 159284, Pittsburgh, Pennsylvania
  - Rhode Island Hospital /ID# 160834, Providence, Rhode Island
  - Sarah Cannon Research Institute-Chattanooga /ID# 202933, Chattanooga, Tennessee
  - Thompson Cancer Survival Ctr /ID# 202460, Knoxville, Tennessee
  - Tennessee Oncology-Nashville Centennial /ID# 161168, Nashville, Tennessee
  - Univ Medical Ctr Brackenridge /ID# 155798, Austin, Texas
  - Parkland Health and Hosp Syste /ID# 170933, Dallas, Texas
  - UT Southwestern Medical Center /ID# 157848, Dallas, Texas
  - Houston Methodist Hospital - Scurlock Tower /ID# 202323, Houston, Texas
  - Medical Oncology Associates /ID# 156715, Spokane, Washington
  - West Virginia Univ School Med /ID# 156687, Morgantown, West Virginia
- Australia (7):
  - Coffs Harbour Hospital /ID# 158880, Coffs Harbour, New South Wales
  - Gosford Hospital /ID# 158884, Gosford, New South Wales
  - Newcastle Private Hospital /ID# 203506, Lambton Heights, New South Wales
  - Royal North Shore Hospital /ID# 158881, Saint Leonards, New South Wales
  - Calvary North Adelaide Hospita /ID# 161701, Adelaide, South Australia
  - Sunshine Hospital /ID# 161700, St Albans, Victoria
  - Affinity Clinical Research Ser /ID# 158887, Nedlands
- Austria (5):
  - SMZ Baumgartner Höhe, Otto-Wagner-Spital und Pflegezentrum /ID# 201776, Vienna, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf /ID# 201768, Vienna, Vienna
  - LKH-Univ. Klinikum Graz /ID# 159563, Graz
  - Ordensklinikum Linz GmbH, Elisabethinen /ID# 159564, Linz
  - Salzburger Landeskliniken (SALK) /ID# 201779, Salzburg
- Belarus (3):
  - Bobruysk Interdistrict Onco. /ID# 169393, Babruysk
  - State Institution Republican Scientific Practical Center of Oncology and Medica /ID# 159383, Lesnoy
  - Mogilev Reg Clin Oncology Dis /ID# 159384, Mogilev
- Belgium (5):
  - CHU Saint-Pierre /ID# 159009, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi /ID# 159006, Charleroi, Hainaut
  - ZNA Middelheim /ID# 159007, Antwerp
  - Hopital de Jolimont /ID# 159005, Haine-Saint-Paul
  - CHU Charleroi (Vesale) /ID# 159008, Montigny-le-Tilleul
- Brazil (8):
  - Hospital Evangelico de Cachoei /ID# 159657, Cachoeiro de Itapemirim, Espírito Santo
  - Liga Norte Rio Grandense Cont. /ID# 159011, Natal, Rio Grande do Norte
  - Associação Hospital de Caridade Ijuí - Centro de Tratamento de Cancer - CACON /ID# 159013, Ijuí, Rio Grande do Sul
  - Associação Hospital Beneficente São Vicente de Paulo - Hospital São Vicente de P /ID# 159661, Passo Fundo, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS /ID# 159662, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos /ID# 159012, Barretos, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto /ID# 159659, São José do Rio Preto, São Paulo
  - Instituto Nacional de Câncer José de Alencar Gomes da Silva (INCA) /ID# 159658, Rio de Janeiro
- Bulgaria (2):
  - UMHAT Tsaritsa Joanna - ISUL /ID# 159638, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 159639, Sofia
- Canada (6):
  - British Columbia Cancer Agency /ID# 163721, Surrey, British Columbia
  - Brampton Civic Hospital /ID# 204425, Brampton, Ontario
  - R.S. McLaughlin Durham Regional /ID# 170870, Oshawa, Ontario
  - Princess Margaret /ID# 170868, Toronto, Ontario
  - Windsor Regional Cancer Centre /ID# 170869, Windsor, Ontario
  - Iucpq-Ul /Id# 159530, Québec, Quebec
- China (13):
  - Fujian Provincial Cancer Hospital /ID# 204864, Fuzhou, Fujian
  - Harbin Medical University Cancer Hospital /Id# 203638, Harbin, Heilongjiang
  - Hubei Cancer Hospital /ID# 202886, Wuhan, Hubei
  - Jilin Cancer Hosptial /ID# 204060, Changchun, Jilin
  - The Affiliated Cancer Hospital of Xinjiang Medical university /ID# 203641, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital /ID# 204911, Kunming, Yunnan
  - Zhejiang Cancer hospital /ID# 204640, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital /ID# 206802, Jianggan Hangzhou, Zhejiang
  - Jiangsu Province Hospital /ID# 205183, Nanjing
  - 4th Military Medical Universit /ID# 203986, Xi'an
  - First Affiliated Hospital of Xi'an Jiaotong University /ID# 203733, Xi'an
  - Henan Cancer Hospital /ID# 203983, Zhengzhou Henan
  - Henan Cancer Hospital /ID# 204636, Zhengzhou Henan
- Croatia (3):
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 159090, Zagreb, City of Zagreb
  - Klinika za plucne bolesti Jordanovac /ID# 159505, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Rijeka /ID# 159504, Rijeka, Primorje-Gorski Kotar County
- Czechia (6):
  - Thomayerova nemocnice /ID# 159062, Prague, Praha 4
  - Nemocnice Rudolfa a Stefanie /ID# 159655, Benešov
  - Nemocnice Horovice a.s. /ID# 161186, Hořovice
  - Vitkovicka nemocnice a. s. /ID# 161187, Ostrava
  - FN Plzen /ID# 204097, Pilsen
  - Oblastni Nemocnice Pribram /ID# 159654, Příbram
- Denmark (4):
  - Rigshospitalet /ID# 158055, Copenhagen Ø, Capital Region
  - Herlev Hospital /ID# 158053, Herlev, Capital Region
  - Aalborg University Hospital /ID# 203737, Aalborg, North Denmark
  - Odense Universitets Hospital /ID# 158054, Odense C, Region Syddanmark
- Estonia (2):
  - East Tallinn Central Hospital /ID# 160019, Tallinn
  - North Estonian Medical Centre /ID# 159779, Tallinn
- Docrates Cancer Center /ID# 159591, Helsinki, Finland
- France (10):
  - CHU Hopital Nord /ID# 160543, Marseille, Bouches-du-Rhone
  - Hopital Haut-Lévêque /ID# 160547, Pessac, Gironde
  - CHU Calmette /ID# 202706, Lille, Hauts-de-France
  - Centre Leon Berard /ID# 160550, Lyon, Rhone
  - Centre Hosp Intercommunal de Creteil /ID# 162686, Créteil, Val-de-Marne
  - Hopital Tenon /ID# 160541, Paris
  - Hospital Pontchaillou /ID# 160544, Rennes
  - Nouvel Hopital Civil (NHC) /ID# 204427, Strasbourg
  - Hopital Larrey /ID# 204290, Toulouse
  - Institut Curie /ID# 207514, Paris, Île-de-France Region
- Germany (9):
  - KH Martha-Maria Halle Dolau /ID# 158794, Halle, Saxony-Anhalt
  - Charite Universitatsmedizin Berlin Campus Virchow Klinikum /ID# 158783, Berlin
  - Evangelische Lungenklinik Berl /ID# 158935, Berlin
  - Asklepios Fachkliniken M. Gaut /ID# 158789, Gauting
  - Thoraxklinik Heidelberg gGmbH /ID# 158871, Heidelberg
  - Lungenklinik Hemer /ID# 158790, Hemer
  - Klinikum Kassel /ID# 158786, Kassel
  - Klinik Loewenstein GmbH /ID# 158870, Löwenstein
  - Fachkliniken Wangen /ID# 160779, Wangen
- Greece (7):
  - Metropolitan General Hospital /ID# 202422, Cholargós, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 159160, Athens
  - Metropolitan Hospital /ID# 159157, Athens
  - University General Hospital of Heraklion PA.G.N.I /ID# 202409, Heraklion
  - University Hospital of Ioannin /ID# 159158, Ioannina
  - General Oncological Hospital /ID# 159159, Nea Kifissia
  - Euromedica General Clinic /ID# 159156, Thessaloniki
- Hong Kong (3):
  - Queen Elizabeth Hospital /ID# 159565, Kowloon
  - Princess Margaret Hospital /ID# 162810, Lai Chi Kok
  - Tuen Mun Hospital /ID# 162435, Tuenmen
- Hungary (5):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 158962, Miskolc, Borsod-Abauj Zemplen county
  - Orszagos Koranyi Pulmonologiai Intezet /ID# 158953, Budapest XII, Budapest
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz - Pulmonologia /ID# 202466, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem /ID# 158955, Budapest
  - Csongrad Megyei Mellkasi Beteg /ID# 158952, Deszk
- Ireland (6):
  - St. James's Hospital /ID# 159712, Dublin, Dublin
  - Cork University Hospital /ID# 159715, Cork
  - St Vincent's University Hosp /ID# 161678, Dublin
  - Beaumont Hospital /ID# 159711, Dublin
  - University Hospital Limerick /ID# 159714, Limerick
  - University Hospital Waterford /ID# 159713, Waterford
- Israel (8):
  - Rabin Medical Center /ID# 159764, Petakh Tikva, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 161467, Tel Aviv, Tel Aviv
  - Soroka University Medical Center /ID# 159762, Beersheba
  - Assaf Harofeh Medical Center /ID# 201883, Be’er Ya‘aqov
  - Rambam Health Care Campus /ID# 202336, Haifa
  - Hadassah /ID# 159763, Jerusalem
  - Meir Medical Center /ID# 159761, Kfar Saba
  - Sheba Medical Center /ID# 159760, Ramat Gan
- Italy (6):
  - IRST IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori /ID# 160898, Meldola, Emilia-Romagna
  - Policlinico Universitario Campus Bio-Medico /ID# 160874, Rome, Lazio
  - AUSL 8 Arezzo Ospedale San Don /ID# 160897, Arezzo
  - A.O.U. San Luigi Gonzaga /ID# 158916, Orbassano
  - Ospedale Santa Maria delle Cro /ID# 158911, Ravenna
  - IFO Istituto Nazionale Tumori /ID# 158912, Rome
- Japan (22):
  - Aichi Cancer Center Hospital /ID# 164976, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 165721, Kashiwa-shi, Chiba
  - Kyushu University Hospital /ID# 165722, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 164595, Kurume-shi, Fukuoka
  - Kanazawa University Hospital /ID# 165127, Kanazawa, Ishikawa-ken
  - Kanagawa Cardiovascular and Respiratory Center /ID# 165015, Yokohama, Kanagawa
  - Yokohama City University Hospital /ID# 165746, Yokohama, Kanagawa
  - Japanese Red Cross Okayama Hospital /ID# 165157, Okayama, Okayama-ken
  - Kansai Medical University Hospital /ID# 165054, Hirakata-shi, Osaka
  - Kindai University Hospital /ID# 166395, Osaka-sayama-shi, Osaka
  - Shizuoka Cancer Center /ID# 166272, Sunto-gun, Shizuoka
  - Tokushima University Hospital /ID# 166105, Tokushima, Tokushima
  - National Cancer Center Hospital /ID# 166547, Chuo-ku, Tokyo
  - Showa University Hospital /ID# 165575, Shinagawa-ku, Tokyo
  - Wakayama Medical University /ID# 165946, Wakayama, Wakayama
  - Hyogo Cancer Center /ID# 165138, Akashi
  - National Hospital Organization Himeji Medical Center /ID# 165899, Himeji
  - Matsusaka City Hospital /ID# 166156, Matsusaka-shi MIE
  - Osaka City General Hospital /ID# 165714, Osaka
  - Hokkaido Cancer Center /ID# 165236, Sapporo
  - Sendai Kousei Hospital /ID# 166491, Sendai
  - Kanagawa Cancer Center /ID# 165814, Yokohama
- Latvia (2):
  - Pauls Stradins Clinical /ID# 158715, Riga
  - Riga East Clinical University /ID# 158716, Riga
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 160016, Kaunas, Kaunas County
  - Klaipeda University Hospital /ID# 160018, Klaipėda
  - National Cancer Institute /ID# 160017, Vilnius
- Mexico (2):
  - Centro de Investigación Clinica Chapultepec /ID# 160965, Morelia, Michoacán
  - Health Pharma professional Ser /ID# 160734, Mexico City
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis /ID# 158081, 's-Hertogenbosch
  - Meander Medisch Centrum /ID# 159064, Amersfoort
  - Rijnstate /ID# 159063, Arnhem
  - Amphia Ziekenhuis /ID# 159065, Breda
  - Catharina Ziekenhuis /ID# 158082, Eindhoven
  - Maastricht Universitair Medisch Centrum /ID# 161669, Maastricht
  - Universitair Medisch Centrum Utrecht /ID# 158083, Utrecht
- Norway (6):
  - Akershus universitetssykehus /ID# 201682, Nordbyhagen, Akershus
  - Drammen Sykehus /ID# 159572, Drammen, Buskerud
  - Haukeland University Hospital /ID# 159573, Bergen, Hordaland
  - St. Olavs Hospital HF /ID# 163110, Trondheim, Sor-Trondelag
  - Radiumhospitalet, OUS /ID# 159574, Oslo
  - Stavanger Universitetssykehus /ID# 159575, Stavanger
- Poland (3):
  - Mrukmed. Lekarz Beata Madej Mruk i Partner /ID# 159604, Rzeszów, Podkarpackie Voivodeship
  - Wojewodzki Szpital Specjalisty /ID# 159603, Bytom
  - Szpitale Pomorskie Sp. z o.o /ID# 159605, Gdynia
- Portugal (7):
  - Centro Hospitalar Lisboa Norte, EPE /ID# 159957, Lisbon, Lisbon District
  - IPO Lisboa FG, EPE /ID# 159949, Lisbon
  - Hospital da Luz, SA /ID# 159954, Lisbon
  - Unidade Local Saude Matosinhos /ID# 159950, Matosinhos Municipality
  - Centro Hospitalar do Porto EPE /ID# 203582, Porto
  - Hospital CUF Porto /ID# 159955, Porto
  - IPO Porto FG, EPE /ID# 159956, Porto
- Russia (11):
  - National Medical Research Cntr /ID# 169885, Moscow, Moscow Oblast
  - Arkhangelsk clinical oncology /ID# 159367, Arkhangelsk
  - Kaluga Regional Clinical Oncol /ID# 160180, Kaluga
  - Clinical Onco Dispensary /ID# 159365, Omsk
  - PMI Euromedservice /ID# 159369, Pushkin
  - LLC Novaya Clinica /ID# 205523, Pyatigorsk
  - LLC BioEq Ltd. /ID# 159368, Saint Petersburg
  - OOO Centre of Palliative Medicine De Vita /ID# 206855, Saint Petersburg
  - N.N. Petrov Research Inst Onc /ID# 159370, Saint Petersburg
  - Ogarev Mordovia State Univ /ID# 205742, Saransk
  - Smolensk Regional Onc Clin Dis /ID# 159372, Smolensk
- Serbia (5):
  - Clinical Center Serbia /ID# 160902, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 160903, Belgrade, Beograd
  - Clinical Center of Nis /ID# 160905, Niš, Nisavski Okrug
  - Institut za onkologiju i radio /ID# 160904, Belgrade
  - Institute For Pulmonary Diseas /ID# 164250, Kamenitz
- South Africa (6):
  - Cancercare Langenhoven Drive Oncology Centre /ID# 159126, Port Elizabeth, Eastern Cape
  - Dr Albert, Bouwer and Jordaan Incorporated /ID# 158873, Pretoria, Gauteng
  - Mary Potter Oncology Centre /ID# 158877, Pretoria, Gauteng
  - The Oncology Centre /ID# 158872, Durban, KwaZulu-Natal
  - Cape Town Oncology Trials /ID# 201311, Cape Town, Western Cape
  - Cancercare Outeniqua Oncology Unit /ID# 200689, George, Western Cape
- South Korea (8):
  - Dong-A University Hospital /ID# 159305, Busan, Busan Gwang Yeogsi
  - CHA Bundang Medical center CHA University /ID# 161281, Seongnam-si, Gyeonggido
  - Kyungpook National University Chilgok Hospital /ID# 159301, Daegu, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 159304, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital /ID# 159302, Seoul, Seoul Teugbyeolsi
  - Chungbuk National University /ID# 159300, Cheongju-si
  - Severance Hospital /ID# 159297, Seoul
  - Asan Medical Center /ID# 159299, Seoul
- Spain (8):
  - Hospital Teresa Herrera - CHUAC /ID# 164368, A Coruña, A Coruna
  - Hospital Regional de Malaga /ID# 164371, Málaga, Malaga
  - Hospital Parc de Salut del Mar /ID# 159690, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 159708, Barcelona
  - Hospital Clinico Universitario San Carlos /ID# 159706, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 159693, Madrid
  - Hospital Universitario La Paz /ID# 159692, Madrid
  - Hospital Clinico Universitario Lozano Blesa /ID# 159709, Zaragoza
- Sweden (5):
  - Centralsjukhuset, Karlstad /ID# 163451, Karlstad, Värmland County
  - Sahlgrenska US Gbg /ID# 159524, Gothenburg, Västra Götaland County
  - University Hospital Linkoping /ID# 159046, Linköping
  - Karolinska Univ Sjukhuset /ID# 159649, Solna
  - Uppsala University Hospital /ID# 159052, Uppsala
- Switzerland (5):
  - Hopitaux Universitaires de Geneve /ID# 160603, Geneva, Canton of Geneva
  - Kantonsspital St. Gallen /ID# 160604, Sankt Gallen, Canton of St. Gallen
  - Universitaetsspital Basel /ID# 160605, Basel
  - Luzerner Kantonsspital /ID# 160607, Lucerne
  - Kantonsspital Winterthur /ID# 161379, Winterthur
- Taiwan (8):
  - China Medical University Hosp /ID# 158981, Taichung, Taichung
  - National Cheng Kung University Hospital /ID# 158799, Tainan, Tainan
  - National Taiwan Univ Hosp /ID# 159049, Taipei City, Taipei
  - Tri-Service General Hospital /ID# 158980, Taipei City, Taipei
  - Dalin Tzu Chi General Hospital /ID# 158983, Dalin Township
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 158798, Kaohsiung City
  - Taichung Veterans General Hosp /ID# 159047, Taichung
  - Taipei Veterans General Hosp /ID# 203699, Taipei
- Turkey (Türkiye) (9):
  - Hacettepe University Medical Faculty /ID# 159242, Altindağ, Ankara
  - Erciyes University Medical Fac /ID# 202269, Melikgazi, Kayseri
  - Ataturk Gogus Hastalikl /ID# 159556, Ankara
  - Akdeniz Universitesi Tip Fakul /ID# 160791, Antalya
  - Bezmi alem Vakif Universitesi /ID# 202267, Istanbul
  - Istanbul Medeniyet Universites /ID# 200126, Istanbul
  - Ege University Medical Faculty /ID# 159243, Izmir
  - Dr. Suat Seren Gogus Has /ID# 159244, Izmir
  - Inonu University /ID# 159245, Malatya
- Ukraine (7):
  - CI Zaporizhzhia Regional Clinical Oncological Dispensary /ID# 159131, Zaporizhzhia, Zaporizhzhia Oblast
  - Regional Municipal Non-Profit Enterprise Bukovynian Clinical Oncology Center /ID# 159864, Chernivtsi
  - Municipal institution Multifie /ID# 159130, Dnipro
  - Regional Center of Oncology /ID# 159132, Kharkiv
  - PE PMC Acinus, Medical and Diagnostic Center /ID# 165543, Kropyvnytskyi
  - Volyn Regional Medical Oncology Centre /ID# 159133, Lutsk
  - Communal Nonprofit Enterprise "Central City Clinical Hospital" of Uzhhorod City /ID# 159865, Uzhhorod
- United Kingdom (11):
  - Cheltenham General Hospital /ID# 169096, Cheltenham, Gloucestershire
  - Queen Elizabeth Medical Centre /ID# 162899, Birmingham
  - The Royal Bournemouth Hospital /ID# 159039, Bournemouth
  - Colchester General Hospital /ID# 159042, Colchester
  - Hereford County Hospital /ID# 159038, Hereford
  - St. George's Healthcare NHS /ID# 202416, London
  - Charing Cross Hospital /ID# 161399, London
  - Maidstone Hospital /ID# 159043, Maidstone
  - Christie NHS Foundation Trust /ID# 159037, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust Freeman Hospital /ID# 159044, Newcastle upon Tyne
  - Torbay Hospital - So Devon HC /ID# 159041, Torquay

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Tanaka K, Isse K, Fujihira T, Takenoyama M, Saunders L, Bheddah S, Nakanishi Y, Okamoto I. Prevalence of Delta-like protein 3 expression in patients with small cell lung cancer. Lung Cancer. 2018 Jan;115:116-120. doi: 10.1016/j.lungcan.2017.11.018. Epub 2017 Nov 22. PMID 29290251

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo every 6 weeks (q6 wk); omitting every third cycle
  Placebo for rovalpituzumab tesirine: Placebo for rovalpituzumab tesirine administered intravenously Day 1 of each 6-week cycle, omitting every third cycle
  Placebo for dexamethasone: Placebo for dexamethasone administered orally twice daily on Day -1, Day 1 (the day of dosing), and Day 2 of each 6 week cycle, omitting every third cycle
- Rovalpituzumab Tesirine/Dexamethasone: Rovalpituzumab tesirine/dexamethasone q6 wk; omitting every third cycle
  Rovalpituzumab tesirine: Rovalpituzumab tesirine 0.3 mg/kg administered intravenously Day 1 of each 6-week cycle, omitting every third cycle
  Dexamethasone: Dexamethasone 8 mg administered orally twice daily on Day -1, Day 1 (the day of dosing), and Day 2 of each 6 week cycle, omitting every third cycle
Period: Overall Study
Arm/Group | Placebo | Rovalpituzumab Tesirine/Dexamethasone
Started | 376 | 372
Completed | 376 | 372
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rovalpituzumab Tesirine/Dexamethasone | Total
Number analyzed (Participants) | 376 | 372 | 748
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.20) | 64.1 (8.40) | 63.9 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 114 | 251
  Male | 239 | 258 | 497
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 15 | 33
  Not Hispanic or Latino | 356 | 355 | 711
  Missing | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 301 | 314 | 615
  Black or African American | 7 | 2 | 9
  Asian | 66 | 55 | 121
  American Indian or Alaska Native | 2 | 0 | 2
  Multiple Races | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With Extensive-Stage Small Cell Lung Cancer With Delta-Like Protein 3 High Expression in Tumor (DLL3high)
Description: OS is defined as the number of months from randomization to death of any cause. Calculated using the Kaplan-Meier methodology.
Time Frame: Survival follow-up continued until the endpoint of death, participant was lost to follow-up or withdrew consent, or termination of the study by AbbVie, whichever occurred first. Median time on study overall was 11.9 months.
Population: DLL3 High Set: all randomized participants with extensive-stage small cell lung cancer with delta-like protein 3 high expression in tumor (DLL3high), defined as ≥ 75% tumor cells staining positive according to the VENTANA DLL3 [SP347] immunohistochemistry [IHC] assay.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Rovalpituzumab Tesirine/Dexamethasone
Number analyzed (Participants) | 240 | 217
months | 9.79 [8.38 to 10.87] | 8.48 [7.26 to 10.18]
Statistical Analysis 1: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Test type: Superiority; p = 0.537, Log Rank — stratified log-rank test; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.84 to 1.36]

2. Secondary Outcome: OS in All Randomized Participants
Description: as for outcome 1
Time Frame: Survival follow-up continued until the endpoint of death, the subject was lost to follow-up or withdrew consent, or termination of the study by AbbVie, whichever occurred first. Median time on study overall was 11.9 months.
Population: Randomized Set: all randomized participants, grouped according to the treatment arm to which they were randomized regardless the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Rovalpituzumab Tesirine/Dexamethasone
Number analyzed (Participants) | 376 | 372
months | 9.89 [8.61 to 11.01] | 8.80 [7.95 to 9.53]
Statistical Analysis 1: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Test type: Superiority; p = 0.237, Log Rank — stratified log-rank test; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.92 to 1.36]

3. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core (EORTC QLQ-C30) Physical Functioning Domain Over Time
Description: The EORTC QLQ-C30 is composed of global health status/QoL scale; five functional domains (physical, role, emotional, cognitive, and social); three symptom domains (fatigue, nausea and vomiting, and pain); and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
  The Physical Functioning domain includes 5 questions in which participants were asked to rate their overall health and overall quality of life as it relates to physical functioning during the past week on a scale from 1 (very poor) to 7 (excellent). The 5 scores were averaged and transformed to a scale from 0 to 100, where a high score represents a high QoL. A positive change from baseline indicates better quality of life.
Time Frame: Baseline, Weeks 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, Final Visit (up to Week 78)
Population: Randomized Set: all randomized participants, grouped according to the treatment arm to which they were randomized regardless the actual treatment received. Participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Rovalpituzumab Tesirine/Dexamethasone
Number analyzed (Participants) | 376 | 372
score on a scale
  Change at Week 6: number analyzed (Participants) | 287 | 296
  Change at Week 6 | -3.97 (1.00) | -4.34 (0.95)
  Change at Week 12: number analyzed (Participants) | 104 | 191
  Change at Week 12 | -1.70 (1.67) | -12.13 (1.27)
  Change at Week 18: number analyzed (Participants) | 9 | 14
  Change at Week 18 | 8.15 (4.02) | -19.52 (4.92)
  Change at Week 24: number analyzed (Participants) | 7 | 11
  Change at Week 24 | -0.95 (7.32) | -19.39 (6.61)
  Change at Week 30: number analyzed (Participants) | 5 | 10
  Change at Week 30 | 5.33 (4.22) | -16.67 (6.78)
  Change at Week 36: number analyzed (Participants) | 2 | 1
  Change at Week 36 | -13.33 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants. | -13.33 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants.
  Change at Week 42: number analyzed (Participants) | 1 | 2
  Change at Week 42 | -6.67 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants. | -3.33 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants.
  Change at Week 48: number analyzed (Participants) | 3 | 2
  Change at Week 48 | -6.67 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants. | -63.33 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants.
  Change at Week 54: number analyzed (Participants) | 1 | 0
  Change at Week 54 | -6.67 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants. |
  Change at Week 60: number analyzed (Participants) | 1 | 1
  Change at Week 60 | 0.00 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants. | 0.00 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants.
  Change at Week 66: number analyzed (Participants) | 2 | 2
  Change at Week 66 | 0.00 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants. | 0.00 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants.
  Change at Week 72: number analyzed (Participants) | 1 | 0
  Change at Week 72 | 0.00 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants. |
  Change at Week 78: number analyzed (Participants) | 1 | 1
  Change at Week 78 | 0.00 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants. | 0.00 (NA) — Statistical model did not support SE estimation for a sample set that was < 5 participants.
  Change at Week Final Visit: number analyzed (Participants) | 298 | 312
  Change at Week Final Visit | -4.14 (1.02) | -13.31 (1.12)
Statistical Analysis 1: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 6; Test type: Superiority; Least Squares (LS) Mean of Difference = -0.36, 95% CI 2-sided [-3.08 to 2.35], Standard Error of Mean 1.39
Statistical Analysis 2: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 12; Test type: Superiority; LS Mean of Difference = -10.43, 95% CI 2-sided [-14.58 to -6.29], Standard Error of Mean 2.12
Statistical Analysis 3: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 18; Test type: Superiority; LS Mean of Difference = -27.67, 95% CI 2-sided [-46.19 to -9.16], Standard Error of Mean 10.57
Statistical Analysis 4: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 24; Test type: Superiority; LS Mean of Difference = -18.44, 95% CI 2-sided [-38.28 to 1.39], Standard Error of Mean 9.99
Statistical Analysis 5: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 30; Test type: Superiority; LS Mean of Difference = -22.00, 95% CI 2-sided [-42.63 to -1.37], Standard Error of Mean 11.27
Statistical Analysis 6: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 36; Test type: Superiority; LS Mean of Difference = 0.00
Statistical Analysis 7: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 42; Test type: Superiority; LS Mean of Difference = 3.33
Statistical Analysis 8: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 48; Test type: Superiority; LS Mean of Difference = -56.67
Statistical Analysis 9: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 60; Test type: Superiority; LS Mean of Difference = 0.00
Statistical Analysis 10: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 66; Test type: Superiority; LS Mean of Difference = -0.00
Statistical Analysis 11: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Week 78; Test type: Superiority; LS Mean of Difference = 0.00
Statistical Analysis 12: Comparison: Placebo vs Rovalpituzumab Tesirine/Dexamethasone; Change at Final Visit; Test type: Superiority; LS Mean of Difference = -9.17, 95% CI 2-sided [-12.16 to -6.19], Standard Error of Mean 1.52

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: participants were followed for survival for a mean of 7.86 months in the Placebo arm and 8.08 months in the Rovalpituzumab Tesirine Plus Dexamethasone arm. Serious and Other Adverse Events: Day 1 of study treatment through 70 days after last treatment. Mean number of weeks on study treatment was 12.8 in the Placebo arm and 17.5 weeks in the Rovalpituzumab Tesirine Plus Dexamethasone arm.
Description: All-Cause Mortality is presented for all participants who were enrolled and randomized. Serious and Other Adverse Events are presented for all participants who were enrolled, randomized, and received at least 1 dose of study medication.
Groups:
- Placebo: Placebo q6 wk; omitting every third cycle
  Placebo for rovalpituzumab tesirine: Placebo for rovalpituzumab tesirine administered intravenously Day 1 of each 6-week cycle, omitting every third cycle
  Placebo for dexamethasone: Placebo for dexamethasone administered orally twice daily on Day -1, Day 1 (the day of dosing), and Day 2 of each 6 week cycle, omitting every third cycle
Arm/Group | Placebo | Rovalpituzumab Tesirine/Dexamethasone
All-Cause Mortality (participants affected / at risk) | 201/376 | 226/372
Serious Adverse Events (participants affected / at risk) | 87/373 | 157/368
Other Adverse Events (participants affected / at risk) | 248/373 | 315/368
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=373) | Rovalpituzumab Tesirine/Dexamethasone (N=368)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 8 (9)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (2)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (2) | 4 (4)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 1 (1) | 0 (0)
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 0 (0) | 1 (1)
EYELID OEDEMA (Eye disorders) | 0 (0) | 1 (1)
PERIORBITAL SWELLING (Eye disorders) | 0 (0) | 2 (2)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 6 (6)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 2 (2)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 3 (4)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 2 (2) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 3 (3)
CHILLS (General disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0)
EUTHANASIA (General disorders) | 1 (1) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 2 (3)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 8 (10) | 9 (11)
GENERALISED OEDEMA (General disorders) | 0 (0) | 2 (2)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 2 (2) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 2 (2) | 2 (2)
SEROSITIS (General disorders) | 0 (0) | 1 (1)
SUDDEN DEATH (General disorders) | 0 (0) | 1 (1)
SWELLING FACE (General disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 2 (2)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 2 (2)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 1 (1)
BILIARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
CORONA VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS CHORIORETINITIS (Infections and infestations) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 2 (2)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
GANGRENE (Infections and infestations) | 0 (0) | 1 (1)
HAEMOPHILUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
KLEBSIELLA INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (3)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
METAPNEUMOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 8 (8) | 14 (16)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 1 (1) | 0 (0)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2) | 6 (8)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 3 (3)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIATION PNEUMONITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD URIC ACID INCREASED (Investigations) | 0 (0) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 3 (4)
OXYGEN SATURATION DECREASED (Investigations) | 1 (1) | 0 (0)
PANCREATIC ENZYMES INCREASED (Investigations) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 1 (2) | 2 (2)
CACHEXIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 (6) | 6 (7)
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (25) | 16 (17)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (10) | 7 (8)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SINONASAL PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BRAIN OEDEMA (Nervous system disorders) | 0 (0) | 1 (1)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2)
DYSMETRIA (Nervous system disorders) | 1 (1) | 0 (0)
EPILEPSY (Nervous system disorders) | 1 (1) | 2 (2)
FACIAL PARESIS (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0)
HYPERAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
PARAPLEGIA (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 1 (1)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 12 (14)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 22 (23)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (11)
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7)
DERMATITIS BULLOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
SHOCK (Vascular disorders) | 0 (0) | 1 (1)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 3 (3) | 2 (2)
VASCULAR COMPRESSION (Vascular disorders) | 1 (1) | 0 (0)
VENA CAVA THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=373) | Rovalpituzumab Tesirine/Dexamethasone (N=368)
ANAEMIA (Blood and lymphatic system disorders) | 11 (18) | 45 (51)
NEUTROPENIA (Blood and lymphatic system disorders) | 10 (11) | 31 (37)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 14 (19) | 61 (79)
PERICARDIAL EFFUSION (Cardiac disorders) | 6 (7) | 58 (63)
ABDOMINAL PAIN (Gastrointestinal disorders) | 14 (14) | 21 (24)
CONSTIPATION (Gastrointestinal disorders) | 35 (37) | 48 (57)
DIARRHOEA (Gastrointestinal disorders) | 35 (39) | 30 (35)
DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 20 (23)
NAUSEA (Gastrointestinal disorders) | 51 (56) | 77 (86)
VOMITING (Gastrointestinal disorders) | 35 (40) | 35 (41)
ASTHENIA (General disorders) | 25 (27) | 34 (48)
FACE OEDEMA (General disorders) | 5 (5) | 41 (48)
FATIGUE (General disorders) | 60 (66) | 91 (112)
OEDEMA PERIPHERAL (General disorders) | 28 (32) | 93 (134)
PYREXIA (General disorders) | 12 (13) | 20 (24)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 (8) | 39 (45)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 12 (13) | 48 (59)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (7) | 29 (44)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 (3) | 19 (21)
WEIGHT DECREASED (Investigations) | 16 (17) | 19 (22)
DECREASED APPETITE (Metabolism and nutrition disorders) | 49 (55) | 95 (115)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (4) | 29 (32)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 3 (4) | 32 (41)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 9 (10) | 27 (34)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 19 (20) | 30 (33)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 29 (29) | 22 (23)
DIZZINESS (Nervous system disorders) | 18 (18) | 30 (34)
HEADACHE (Nervous system disorders) | 19 (19) | 31 (39)
INSOMNIA (Psychiatric disorders) | 13 (13) | 33 (33)
COUGH (Respiratory, thoracic and mediastinal disorders) | 43 (47) | 56 (69)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 39 (41) | 67 (83)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 76 (98)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 23 (27)
DRY SKIN (Skin and subcutaneous tissue disorders) | 9 (9) | 21 (21)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 (6) | 22 (38)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 5 (5) | 88 (128)
PRURITUS (Skin and subcutaneous tissue disorders) | 17 (18) | 21 (25)
RASH (Skin and subcutaneous tissue disorders) | 8 (9) | 24 (30)
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 6 (6) | 22 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (3):
  • Study Protocol (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03033511/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT03033511/SAP_001.pdf
  • Informed Consent Form (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03033511/ICF_002.pdf